CLINICAL TRIAL: NCT04876378
Title: Impact of Breast Cancer Treatment on Joint Health, Cartilage Composition, and Bone Structure in the Knee and Hand
Status: Terminated | Type: Observational
Why Stopped: Funding
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 20923; NCI-2020-03535 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-05-05; First posted 2021-05-06 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Hormone Receptor Positive Breast Adenocarcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diagnostic (questionnaires, MRI): Patients complete a series of questionnaires over 15 minutes about knee function and pain, as well as physical activity. Patients also undergo an MRI over 60 minutes.
  Interventions: Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study investigates the impact of breast cancer treatment on joint health, cartilage, composition, and bone structure in the knee and hand in patients with hormone-receptor positive stage I-III breast cancer and healthy patients. The investigators will use Magnetic Resonance Imaging (MRI) to assess the quality of hand and knee joints. This study may help doctors learn more about hand and knee joint pain that occurs during aromatase inhibitor treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate pathological alterations in cartilage and joints in breast cancer patients on aromatase inhibitor (AI)s with and without pain and in healthy control patients.

OUTLINE:

Patients complete a series of questionnaires over 15 minutes about knee function and pain, as well as physical activity. Patients also undergo an MRI of about 60 minutes.

After completion of study, a subset of patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from participant or participant's legal representative and ability for participant to comply with the requirements of the study
2. Breast cancer patients with either natural or chemically induced menopause with stage 1-3 hormone receptor-positive breast cancers and on AI for at least one year OR healthy postmenopausal women

   Breast cancer patients on aromatase inhibitors (AI) may fall into one of the three following groups:
   * Patients with knee pain with Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) >= 5, but no or minimal hand/wrist pain
   * Patients with self-reported moderate or severe hand/wrist pain but no or only mild knee pain (WOMAC =< 7)
   * Patients with no or minimal hand/wrist or knee pain (WOMAC =< 7)
3. Age <= 70 years old
4. Ability to read and complete quality of life surveys in English (or have a family member or friend available to translate and assist in completing surveys)

Exclusion Criteria:

1. History of prior traumatic injury at knee joint or severe degenerative joint disease or osteoarthritis defined as having a history of prior joint replacement or moderate to severe knee pain prior to initiation of AI
2. History of claustrophobia
3. Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data, including prior history of implanted devices with ferromagnetic objects

Max Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of breast cancer and normal controls.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Mean differences in hyaline cartilage biochemical composition | Up to 6 months
  Will determine differences in hyaline cartilage biochemical composition (using magnetic resonance imaging) between breast cancer patients under aromatase inhibitor (AI) treatment. Linear regression models will be used to assess differences in joint parameters outcomes between healthy controls, AI patients with pain, and AI patients without pain (predictors).
Differences in morphological joint abnormalities | Up to 6 months
  Will determine differences in morphological joint abnormalities (using semi-quantitative magnetic resonance-based scores) between breast cancer patients under aromatase inhibitor (AI) treatment. Linear regression models will be used to assess differences in joint parameters outcomes between healthy controls, AI patients with pain, and AI patients without pain (predictors).

CONTACTS AND LOCATIONS:
Overall Officials: Roland Krug, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No